CLINICAL TRIAL: NCT06172738
Title: The Left Atrial Appendage Closure by Surgery and the Incidence of Stroke in Patients Undergoing Open-heart Surgery Irrespective of Preoperative Atrial Fibrillation Status and Stroke Risk.
Brief Title: The Left Atrial Appendage Closure by Surgery and the Incidence of Stroke in Patients Undergoing Open-heart Surgery.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Beshoy Allam Moris, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Left atrial appendage closure.
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Left Atrial Appendage Thrombosis
Keywords: surgical closure of the left atrial appendage.; stroke; Post operative atrial fibrillation.
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized control trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A. (Experimental): surgical closure of the left atrial appendage.
  Interventions: Procedure: the left atrial appendage closure through surgery.
- group B. (No Intervention): There was no surgical closure of the left atrial appendage.

INTERVENTIONS:
Procedure: the left atrial appendage closure through surgery. — Surgical closure of the left atrial appendage during the set of an elective open heart surgery with the inclusion criteria fulfilled.
  Other Names: LAACS
  Arms: group A.

SUMMARY:
This study aims to assess the efficacy and safety of prophylactic surgical closure of the left atrial appendage for stroke and cardiovascular death prevention in patients undergoing open heart surgery, regardless of their preoperative AF status and stroke risk.

DETAILED DESCRIPTION:
Cerebrovascular complications following cardiac surgical procedures are a significant source of morbidity and mortality. The etiology of postoperative stroke is multifactorial and may include carotid artery stenosis, hypotension, cardiac arrhythmia, aortic atherosclerosis, and transient hypercoagulable state.

Most strokes complicating cardiac surgery occur in patients without significant carotid disease and are acquired after the patient awakens neurologically intact. The high incidence of postoperative AF in these patients suggests a possible embolic cause for some strokes. As such, some postoperative strokes may be preventable.

Previous studies report incident AF in 10 to 65% of patients after open heart surgery, with the highest incidences after a combination of coronary artery bypass grafting (CABG) and valve surgery.

In patients with non-operative AF, the risk of ischemic stroke is markedly reduced by adequate OAC. However, the management of postoperative AF is still a challenge and is, by some, regarded as a transient phenomenon not requiring intervention. The risk of bleeding poses a significant limitation to the use of OAC, which consequently increases focus on left atrial appendage (LAA) closure, as the LAA is a predilection site for thrombus formation during AF.

Based on previous studies, ≥90% of AF-related left atrial thrombi are located in the left atrial appendage (LAA), and therefore, LAA occlusion is a tempting method for AF-related stroke prevention.

Current recommendations regarding surgical left atrial appendage (LAA) closure to prevent thromboembolisms lack high-level evidence.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years scheduled for first-time planned open-heart surgery.

Exclusion Criteria:

Pediatric population >18 years. Emergent open heart surgery. Patients with current endocarditis. Where follow-up is not possible. The patient refused to sign the informed consent to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Stroke. | 2 years post operative.
  the incidence of stroke in patients undergoing open-heart surgery, including transient ischemic attack, as assigned by two independent neurologists blinded to the treatment allocation.
Mortality | 2 years post operative.
  post-operative mortality rate.

SECONDARY OUTCOMES:
Postoperative arrhythmias. | 1 year
  Incidence of postoperative arrhythmias with special regard to post-operative AF.
Hospital stay. | 1 month
  Number of inpatient hospital stay days.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li Y, Walicki D, Mathiesen C, Jenny D, Li Q, Isayev Y, Reed JF 3rd, Castaldo JE. Strokes after cardiac surgery and relationship to carotid stenosis. Arch Neurol. 2009 Sep;66(9):1091-6. doi: 10.1001/archneurol.2009.114. PMID 19752298
- [Background] Murdock DK, Rengel LR, Schlund A, Olson KJ, Kaliebe JW, Johnkoski JA, Riveron FA. Stroke and atrial fibrillation following cardiac surgery. WMJ. 2003;102(4):26-30. PMID 12967018
- [Background] Park-Hansen J, Holme SJV, Irmukhamedov A, Carranza CL, Greve AM, Al-Farra G, Riis RGC, Nilsson B, Clausen JSR, Norskov AS, Kruuse CR, Rostrup E, Dominguez H. Adding left atrial appendage closure to open heart surgery provides protection from ischemic brain injury six years after surgery independently of atrial fibrillation history: the LAACS randomized study. J Cardiothorac Surg. 2018 May 23;13(1):53. doi: 10.1186/s13019-018-0740-7. PMID 29792215
- [Background] Kiviniemi T, Bustamante-Munguira J, Olsson C, Jeppsson A, Halfwerk FR, Hartikainen J, Suwalski P, Zindovic I, Copa GR, van Schaagen FRN, Hanke T, Cebotari S, Malmberg M, Fernandez-Gutierrez M, Bjurbom M, Schersten H, Speekenbrink R, Riekkinen T, Ek D, Vasankari T, Lip GYH, Airaksinen KEJ, van Putte B; LAA-CLOSURE Investigators. A randomized prospective multicenter trial for stroke prevention by prophylactic surgical closure of the left atrial appendage in patients undergoing bioprosthetic aortic valve surgery--LAA-CLOSURE trial protocol. Am Heart J. 2021 Jul;237:127-134. doi: 10.1016/j.ahj.2021.03.014. Epub 2021 Mar 30. PMID 33798494
- [Background] Madsen CL, Park-Hansen J, Irmukhamedov A, Carranza CL, Rafiq S, Rodriguez-Lecoq R, Palmer-Camino N, Modrau IS, Hansson EC, Jeppsson A, Hadad R, Moya-Mitjans A, Greve AM, Christensen R, Carstensen HG, Host NB, Dixen U, Torp-Pedersen C, Kober L, Gogenur I, Truelsen TC, Kruuse C, Sajadieh A, Dominguez H; LAACS-2 trial Investigators. The left atrial appendage closure by surgery-2 (LAACS-2) trial protocol rationale and design of a randomized multicenter trial investigating if left atrial appendage closure prevents stroke in patients undergoing open-heart surgery irrespective of preoperative atrial fibrillation status and stroke risk. Am Heart J. 2023 Oct;264:133-142. doi: 10.1016/j.ahj.2023.06.003. Epub 2023 Jun 10. PMID 37302738